CLINICAL TRIAL: NCT06709183
Title: The Effect of Oral Care Retractor Developed for Intubated Patients in Intensive Care Unit on Oral Care Practices
Brief Title: Oral Care Apparatus for Intubated Patients
Acronym: Oral Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Hasret Topalı, PhD student, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2024Phd
Record Dates: First submitted 2024-11-20; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Intensive Care; Oral Care; Intubated ICU Patients
Keywords: intensive care; oral care; oral care retractor; intubated ICU patients

STUDY DESIGN:
Intervention Model Description: The research will be conducted through simulation using a standard mannequin in room 428 in the general intensive care unit. Room 428 in the general intensive care unit is a standard intensive care room with four walls of glass, 15 m2 in size, one supply cabinet, one cloakroom, oxygen panel, mechanical ventilator, monitor and single bed, where patients can be monitored instantly with a camera system. In our study, this intensive care room will be used to evaluate the effectiveness of the oral care retractor designed for intensive care patients in order to ensure that oral care procedures to be applied by nurses are in a realistic environment and that nurses feel as if they are applying to a live patient.
  Simulation method will be used for the experimental study part of this research. Laerdal brand MegaCode Kelly emergency care simulator will be used in the study.
Masking Description: Assistant researcher
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Standard oral care (Control - intervention) (Sham Comparator): The nurses in the control-intervention group will perform standard oral care in the first oral care and oral care using the oral care retractor in the second oral care.
  Interventions: Other: Control - intervention
- Oral care retractor (Intervention - Control) (Active Comparator): The nurses in the intervention-control group will perform the first oral care with an oral care retractor, and in the second oral care, they will perform standard oral care without using an oral care retractor.
  Interventions: Other: Intervention-Control

INTERVENTIONS:
Other: Intervention-Control — Nurses in this group will start the first oral care practice by using the oral care retractor on the model. Before starting the procedure, the nurses will fill in the 'Beck Mouth Assessment Guide' and after the procedure, they will fill in the 'Oral Care Practices Evaluation Form'. A rest period of at least 10 minutes will be provided before the second oral care application. Standard oral care will be applied during the second application. Similarly, nurses will complete the 'Beck Oral Assessment Guide' before the procedure and the 'Oral Care Practices Assessment Form' after the procedure. At the end of both procedures, nurses will complete the 'Quebec Assistive Technology User Satisfaction Assessment Questionnaire (Q-ATUSA)' and the 'Interview Form'. The 'Interview Form' will be used to collect nurses' experiences and opinions about the oral care procedure. During the interview, audio recordings will be made with the knowledge of the nurses.
  Other Names: Oral care retractor
  Arms: Oral care retractor (Intervention - Control)
Other: Control - intervention — In the first oral care procedure, nurses in this group will perform standard oral care on the model without using the oral care retractor. They will complete the 'Beck Oral Assessment Guide' before the procedure and the 'Oral Care Practices Evaluation Form' after the procedure. There will be a rest period of at least 10 minutes before the second oral care procedure. During this procedure, the second group of nurses who initially perform standard oral care will perform oral care using an oral care retractor. Similarly, they will complete the 'Beck Oral Assessment Guide' before the procedure and the 'Oral Care Practices Evaluation Form' after the procedure. At the end of both procedures, nurses will complete the 'Quebec Assistive Technology User Satisfaction Assessment Questionnaire (Q-ATUSA)' and the 'Interview Form'. The 'Interview Form' will be used to obtain nurses' experiences and opinions regarding oral care practices..
  Other Names: Standard oral care
  Arms: Standard oral care (Control - intervention)

SUMMARY:
There are several practical challenges in providing oral care to intubated patients. The presence of an endotracheal tube often makes it difficult to thoroughly evaluate the oral cavity, and there is a risk of tube displacement or removal during oral care. Additionally, the lack of standardized care protocols, limited time, and inadequate equipment further complicate the assessment of oral mucosal membranes, increase the likelihood of complications, and prolong ICU stays. The literature also highlights that intubated patients often exhibit behaviors such as gagging, biting the tube, or turning their head during oral care. These actions make it challenging for ICU nurses to use oral care tools effectively, resulting in insufficient evaluation and cleaning of the oral cavity. In a study conducted by Dale et al., ICU healthcare workers emphasized the need for an oral device that could withstand biting pressure, keep the teeth separated, and be flexible enough to prevent discomfort while enabling effective oral care. However, the literature does not report the existence of a device designed to open the oral cavity for intubated patients during oral care. Inspired by cheek retractors used in dentistry, this project aims to design an oral care retractor specifically for intubated patients. This device would facilitate the evaluation of the oral cavity and provide a clear view during oral care, enabling effective oral hygiene practices.

DETAILED DESCRIPTION:
Intensive care units (ICUs) are facilities where basic and advanced life support are provided for patients who are completely bedridden, unable to perform daily living activities, and require constant nursing care. These patients often receive oxygen therapy or mechanical ventilation. Most ICU patients are dependent on nursing care, placing significant responsibilities on ICU nurses to meet self-care needs. One of these essential self-care interventions is oral care.

Oral care includes approaches such as assessing the oral cavity, maintaining saliva production, preventing the formation of microorganisms, reducing plaque and related diseases, and cleaning and moisturizing oral tissues. Effective oral care provides comfort and helps prevent infections. The absence of regular and effective oral care in ICU patients allows pathogens to proliferate in the oral cavity, increasing microbial load. Patients undergoing endotracheal intubation and mechanical ventilation are particularly at risk for developing systemic infections such as oral infections or healthcare-associated pneumonia. Endotracheal tubes can lead to debris accumulation, create an environment conducive to microbial growth, and keep the mouth continuously open, resulting in xerostomia, dental plaque buildup, and reduced saliva production. Oral care reduces bacterial colonization in the oropharyngeal cavity and prevents adverse outcomes such as poor oral health and respiratory infections.

There are, however, practical challenges in providing oral care to intubated patients. These challenges include difficulty in thoroughly assessing the oral cavity due to the presence of the endotracheal tube, the risk of tube displacement or removal during oral care, the lack of standardized care protocols, and limited time and equipment. These factors complicate the evaluation of oral mucosal membranes, increase the likelihood of complications, and prolong hospital stays. Additionally, the literature notes that intubated patients often exhibit challenging behaviors during oral care, such as gagging, biting the tube, or turning their head, making it difficult for ICU nurses to use oral care tools effectively. This can result in insufficient evaluation and cleaning of the oral cavity. In a study by Dale et al., ICU healthcare workers expressed the need for an oral device that could resist biting pressure, keep the teeth separated, and be flexible enough to prevent discomfort while enabling effective oral care. Inspired by cheek retractors used in dentistry, we designed an oral care retractor to facilitate the evaluation of the oral cavity in intubated patients and enable clear visualization during oral care. This study aims to assess the impact of this newly developed oral care retractor on oral care practices in intubated patients in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Having at least 6 months of work experience in an intensive care unit (Sayın, 2020),
* Working as a nurse in adult intensive care units.

Exclusion Criteria:

* Working as a nurse in a neonatal intensive care unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Effect on oral care applications | It will be filled 2 minutes after the end of the application.
  Whether the oral care retractor has an effect on oral care practices in intubated patients will be evaluated with the Oral Care Practice Evaluation Form. This form was created by the researcher in line with the literature (Dagnew et al., 2020; Dale et al., 2018; Thapa & Shrestha, 2019) and consists of 4 questions. Nurses will be asked to rate the oral care practice according to the Visual Analogue Scale (VAS) between 0 and 10. VAS ratings will be categorised as low (0-3), medium (4-6) and high (7-10) (Dale et al., 2018).
Oral cavity assessment | It will be filled 2 minutes after the end of the application.
  It will be examined whether the oral care retractor has an effect on the assessment of the oral cavity of intubated patients. Beck oral cavity assessment form will be used for this purpose.This scale was developed by Becks (1979). It has five subscales: lips, gums, oral mucosa, tongue, teeth and saliva, each scored on a four-point Likert scale. The total score of this tool is 5-20. A low score indicates good oral health and a high score indicates the presence of problems. Therefore, 5-10 points indicate mild dysfunction, 11-15 points indicate moderate dysfunction and 16-20 points indicate severe dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Bitlis State Hospital, Bitlis, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayrak-Kahraman, B., Özdemir, L. 2016. "Evaluation of behavioral and physiological pain indicators of intensive care patients during invasive interventions". Journal of Research and Development in Nursing, 18(3), 13-21.
- [Background] Bayrak, S., Akın, S. 2022. "Investigation of intensive care nurses' knowledge and practices regarding oral care interventions applied to intubated patients". Hamidiye University of Health Sciences.
- [Background] Kara, A., Bölükbaş, N. 2019. "Determination of pain behaviors in intubated intensive care patients with endotracheal tube and oral care". Ordu University.
- [Background] Korhan, E. A., Yönt, G. H., Demiray, A., Akça, A., Eker, A. 2015. "Determination of nursing diagnoses in intensive care unit and evaluation according to Nanda diagnoses". 5(1), 16-21.
- [Background] Özdemir, S. 2020. "The effect of different concentrations of chlorhexidine used in oral care of patients on mechanical ventilation support on microbial colonization". Aydın Adnan Menderes University.
- [Background] Yakut E, Duger T, Oksuz C, Yorukan S, Ureten K, Turan D, Frat T, Kiraz S, Krd N, Kayhan H, Yakut Y, Guler C. Validation of the Turkish version of the Oswestry Disability Index for patients with low back pain. Spine (Phila Pa 1976). 2004 Mar 1;29(5):581-5; discussion 585. doi: 10.1097/01.brs.0000113869.13209.03. PMID 15129077
- [Background] Yildiz M, Durna Z, Akin S. Assessment of oral care needs of patients treated at the intensive care unit. J Clin Nurs. 2013 Oct;22(19-20):2734-47. doi: 10.1111/jocn.12035. Epub 2013 Mar 27. PMID 23534462
- [Background] Vollman, K., Sole, M. Lou, Quinn, B. 2017. "Endotracheal tube care and oral care practices for ventilated and non-ventilated patients". In Procedure Manual for High Acuity, Progressive, and Critical Care (pp. 32-39).
- [Background] Thapa, B., Shrestha, R. 2019. "Nurses' knowledge and practice regarding oral care in intubated patients at selected teaching hospitals, Chitwan". International Journal of Innovative Science and Research Technology, 4(5).
- [Background] Terzi, B., Kaya, N. 2011. "Nursing care of critically ill patients". Yoğun Bakım Dergisi.
- [Background] Terezakis E, Needleman I, Kumar N, Moles D, Agudo E. The impact of hospitalization on oral health: a systematic review. J Clin Periodontol. 2011 Jul;38(7):628-36. doi: 10.1111/j.1600-051X.2011.01727.x. Epub 2011 Apr 7. PMID 21470276
- [Background] Sachdev M, Ready D, Brealey D, Ryu J, Bercades G, Nagle J, Borja-Boluda S, Agudo E, Petrie A, Suvan J, Donos N, Singer M, Needleman I. Changes in dental plaque following hospitalisation in a critical care unit: an observational study. Crit Care. 2013 Sep 4;17(5):R189. doi: 10.1186/cc12878. PMID 24007571
- [Background] Prendergast V, Kleiman C, King M. The Bedside Oral Exam and the Barrow Oral Care Protocol: translating evidence-based oral care into practice. Intensive Crit Care Nurs. 2013 Oct;29(5):282-90. doi: 10.1016/j.iccn.2013.04.001. Epub 2013 May 20. PMID 23702324
- [Background] Noddeskou LH, Hemmingsen LE, Hordam B. Elderly patients' and nurses' assessment of traditional bed bath compared to prepacked single units--randomised controlled trial. Scand J Caring Sci. 2015 Jun;29(2):347-52. doi: 10.1111/scs.12170. Epub 2014 Sep 6. PMID 25196742
- [Background] Miura K, Kadone H, Abe T, Koda M, Funayama T, Noguchi H, Kumagai H, Nagashima K, Mataki K, Shibao Y, Sato K, Kawamoto H, Sankai Y, Yamazaki M. Successful Use of the Hybrid Assistive Limb for Care Support to Reduce Lumbar Load in a Simulated Patient Transfer. Asian Spine J. 2021 Feb;15(1):40-45. doi: 10.31616/asj.2019.0111. Epub 2020 Feb 4. PMID 32008308
- [Background] Kumsar, A. K., Yilmaz, F. T. 2013. "The effects of intensive care units on critically-ill patients and nursing care". Journal of Education and Research in Nursing, 10(2), 56-61.
- [Background] Jansson MM, Syrjala HP, Ohtonen PP, Merilainen MH, Kyngas HA, Ala-Kokko TI. Effects of simulation education on oral care practices - a randomized controlled trial. Nurs Crit Care. 2017 May;22(3):161-168. doi: 10.1111/nicc.12276. Epub 2017 Jan 16. PMID 28093837
- [Background] Jang CS, Shin YS. Effects of combination oral care on oral health, dry mouth and salivary pH of intubated patients: A randomized controlled trial. Int J Nurs Pract. 2016 Oct;22(5):503-511. doi: 10.1111/ijn.12460. Epub 2016 Jun 28. PMID 27349717
- [Background] Hua, B., Mu, R., Shi, H., Inniss, E., Yang, J. 2016. "Water quality in selected small drinking water systems of missouri rural communities". Beverages 2016, Vol. 2, Page 10, 2(2), 10.
- [Background] Dale CM, Smith O, Burry L, Rose L. Prevalence and predictors of difficulty accessing the mouths of intubated critically ill adults to deliver oral care: An observational study. Int J Nurs Stud. 2018 Apr;80:36-40. doi: 10.1016/j.ijnurstu.2017.12.009. Epub 2017 Dec 28. PMID 29353710
- [Background] Dale CM, Angus JE, Sutherland S, Dev S, Rose L. Exploration of difficulty accessing the mouths of intubated and mechanically ventilated adults for oral care: A video and photographic elicitation study. J Clin Nurs. 2020 Jun;29(11-12):1920-1932. doi: 10.1111/jocn.15014. Epub 2019 Aug 20. PMID 31342565
- [Background] Dagnew ZA, Abraham IA, Beraki GG, Mittler S, Achila OO, Tesfamariam EH. Do nurses have barriers to quality oral care practice at a generalized hospital care in Asmara, Eritrea? A cross-sectional study. BMC Oral Health. 2020 May 20;20(1):149. doi: 10.1186/s12903-020-01138-y. PMID 32434570
- [Background] Croft K, Dallal-York J, Miller S, Anderson A, Donohue C, Jeng E, Plowman EK. Provision of Oral Care in the Cardiothoracic Intensive Care Unit: Survey of Nursing Staff Training, Confidence, Methods, Attitudes, and Perceived Barriers. J Contin Educ Nurs. 2023 Jul;54(7):313-321. doi: 10.3928/00220124-20230620-02. Epub 2023 Jul 1. PMID 37390307
- [Background] Choi MI, Noh HJ, Han SY, Bae SS, Kim G, Mun SJ. Development and evaluation of simulation-based scenario education program for professional oral hygiene care in intubated patient. J Dent Educ. 2023 Nov;87(11):1512-1522. doi: 10.1002/jdd.13345. Epub 2023 Aug 2. PMID 37530076
- [Background] Cecon F, Ferreira LE, Rosa RT, Gursky LC, de Paula e Carvalho A, Samaranayake LP, Rosa EA. Time-related increase of staphylococci, Enterobacteriaceae and yeasts in the oral cavities of comatose patients. J Microbiol Immunol Infect. 2010 Dec;43(6):457-63. doi: 10.1016/S1684-1182(10)60071-0. PMID 21195971
- [Background] Blot, S., Vandijck, D., Labeau, S. 2008. "Oral care of intubated patients". Clinical Pulmonary Medicine, 15, 153-160.
- [Background] Batiha, A.-M., Alhalaiqa, F. N., Bashayreh, I., Saifan, A., Al-Zaru, I. M., Omran, S. 2015. "Comprehensive Oral Care Program for Intubated Intensive Care Unit Patients". Advanced Studies in Biology, 7(6), 259-273.
- [Background] Al-Zaru, I. M., Batiha, A. M., Al-Talla, A. A., Bani, Y. M., Alhalaiqa, F. N. 2020. "Knowledge, attitudes, and practices of oral care in mechanical ventilated patients". Prakticky Lekar, 100(January), 5-11.
- [Background] Andersson M, Wilde-Larsson B, Persenius M. Intensive care nurses fail to translate knowledge and skills into practice - A mixed-methods study on perceptions of oral care. Intensive Crit Care Nurs. 2019 Jun;52:51-60. doi: 10.1016/j.iccn.2018.09.006. Epub 2018 Oct 5. PMID 30297151